CLINICAL TRIAL: NCT05152927
Title: Evaluating Impact of Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Parathyroidectomy
Brief Title: Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Parathyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21208; 5R01CA212147-02 (NIH)
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Parathyroid Diseases; Parathyroid Dysfunction; Parathyroid Neoplasms; Parathyroid Adenoma; Hypercalcemia; Neoplasms, Glandular and Epithelial; Endocrine Gland Neoplasms; Adenoma; Hyperparathyroidism; Hyperparathyroidism, Primary
Keywords: Near Infrared Autofluorescence; Parathyroidectomy; Intraoperative Parathyroid Identification; Persistent Hyperparathyroidism; Persistent Hypercalcemia; Failed Parathyroidectomy; Repeat Parathyroidectomy
MeSH Terms: conditions — Parathyroid Diseases; Parathyroid Neoplasms; Hypercalcemia; Neoplasms, Glandular and Epithelial; Endocrine Gland Neoplasms; Adenoma; Hyperparathyroidism; Hyperparathyroidism, Primary

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only participants will be masked to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Parathyroid Eye (PTeye) (Experimental): For patients assigned to the study arm, the surgeon will use the PTeye as an intraoperative tool to identify if a suspect tissue is a parathyroid or not, during the parathyroid surgery.
  Interventions: Device: Parathyroid Eye (PTeye)
- Usual Standard of Care (No Intervention): The surgeon will proceed with the parathyroid surgery as usual, while relying solely on her/his surgical experience in identifying the parathyroid glands during the operations.

INTERVENTIONS:
Device: Parathyroid Eye (PTeye) — Intraoperative Tool
  Other Names: Near Infrared Autofluorescence (NIRAF); NIRAF detection modality; PTeye
  Arms: Parathyroid Eye (PTeye)

SUMMARY:
The goal of this study is to assess whether using PTeye (AiBiomed, Santa Barbara, CA) - a NIRAF detection modality - can improve patient outcomes and reduce healthcare associated costs after parathyroid surgeries. By being able to quickly and definitively locate parathyroid glands while in the operating room, the duration of surgical procedure could be further reduced. In addition, the number of frozen section biopsy and associated costs can be minimized. Furthermore, repeat surgeries as a result of missing a diseased parathyroid gland at the time of the initial parathyroidectomy for hyperparathyroidism could potentially be avoided.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, randomized study comparing the use of PTeye during parathyroidectomy to usual standard practice.

PRIMARY OBJECTIVES:

I. Assess the impact of PTeye on intra-operative identification of parathyroid tissues.

II. Assess the impact of PTeye on improving efficiency of parathyroid surgeries.

III. Assess the impact of PTeye on minimizing risk of post-surgical complications.

Participants will be randomized to either the experimental or control arm.

The surgeon will first take 5 baseline NIRAF measurements on the thyroid gland (or neck muscles, if thyroid is absent) using the disposable sterile fiber probe that is connected to the PTeye console, as per device functionality requirements. The subsequent step would involve touching the target tissue in the neck with the fiber optic probe, following which the PTeye will indicate to the surgeon if the tissue is likely parathyroid or not.

For patients assigned to the control arm, the surgeon will not use the PTeye and will proceed with the parathyroid surgery as usual, while relying solely on her/his surgical experience in identifying the parathyroid glands during the operations.

Participants will be follow-ed up for up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adults >=18 years old) patients with primary hyperparathyroidism who will be undergoing parathyroid surgery
* All adult (>=18 years old) patients with persistent primary hyperparathyroidism after having undergone a failed prior parathyroid surgery who will be undergoing repeat parathyroid surgery

Exclusion Criteria:

* Children and minors
* Pregnant women
* Patients with concurrent parathyroid and thyroid disease that require total thyroidectomy
* Patients with secondary or tertiary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quan-Yang Duh, MD, FACS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McWade MA, Paras C, White LM, Phay JE, Mahadevan-Jansen A, Broome JT. A novel optical approach to intraoperative detection of parathyroid glands. Surgery. 2013 Dec;154(6):1371-7; discussion 1377. doi: 10.1016/j.surg.2013.06.046. PMID 24238054
- [Background] Thomas G, Solorzano CC, Baregamian N, Mannoh EA, Gautam R, Irlmeier RT, Ye F, Nelson JA, Long SE, Gauger PG, Magner A, Metcalf T, Shirley LA, Phay JE, Mahadevan-Jansen A. Comparing intraoperative parathyroid identification based on surgeon experience versus near infrared autofluorescence detection - A surgeon-blinded multi-centric study. Am J Surg. 2021 Nov;222(5):944-951. doi: 10.1016/j.amjsurg.2021.05.001. Epub 2021 May 13. PMID 34024629
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Groups:
- Parathyroid Eye (PTeye): For participants assigned to the study arm, the surgeon will use the PTeye as an intraoperative tool to identify if a suspect tissue is a parathyroid or not, during the parathyroid surgery.
Period: Overall Study
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Started | 38 | 41
Completed | 38 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Median (Full Range); unit: years] | 68 [25 to 87] | 64 [39 to 81] | 67 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 2 | 4
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Frozen Sections (or Parathyroid Aspirate) Sent for Analysis
Description: Median number of frozen sections (or aspirate) sent for analysis during the parathyroidectomy (PTx) procedure to confirm potential parathyroid tissue
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Measure: Median (Full Range); unit: frozen aspirate samples
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
frozen aspirate samples | 0 [0 to 1] | 0 [0 to 1]

2. Secondary Outcome: Number of Participants With Persistent Hyperparathyroidism (Immediate)
Description: Failure of intra-operative parathyroid hormone (PTH) to normalize (defined as failure of PTH to drop > 50% of its baseline value at final intra-operative PTH assay and/or failure of PTH to drop < 65 pg/ml or 6.9 pmol/L). Participants will be categorized as having persistent hyperparathyroidism (Immediate) Yes or No.
Time Frame: 5-14 days after PTx procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Persistent Hyperparathyroidism or Hypercalcemia (Transient)
Description: Elevated blood calcium levels (total blood calcium level > 10.5 mg/dL or 2.6 mmol/L) with/without elevated parathyroid hormone (PTH) (serum intact PTH > 65 pg/ml or 6.9 pmol/L) at first postoperative visit. Participants will be categorized as having persistent hyperparathyroidism or hypercalcemia (transient) Yes or No.
Time Frame: 5-14 days after PTx procedure
Population: Participants from both groups were missing labs. Not all PTEye participants returned to the clinic for blood draws within 5-14 days to obtain lab values required to calculate this endpoint and standard clinical care does not necessitate participants returning for labs routinely at each follow-up time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 21 | 20
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Persistent Hyperparathyroidism or Hypercalcemia (Failed Parathyroidectomy)
Description: If blood calcium with/without parathyroid hormone (PTH) has not normalized at 1st post-operative visit, calcium and/or PTH is subsequently measured as necessary. Patient is defined to have a failed parathyroidectomy if hypercalcemia/hyperparathyroidism (defined as total blood calcium level > 10.5 mg/dL or 2.6 mmol/L, with/without elevated serum intact PTH > 65 pg/ml or 6.9 pmol/L) persists at or after the 6th postoperative month. Participants will be categorized has having persistent hyperparathyroidism or hypercalcemia (failed parathyroidectomy), Yes or No.
Time Frame: Up to 6 months after PTx procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 29 | 33
Participants | 0 | 1

5. Secondary Outcome: Number of Parathyroid Glands (PG) Identified
Description: Overall number of parathyroid glands identified (Combined both the experimental Group (Glands identified with naked eye + NIRAF) and Control Group (Glands identified with naked eye)
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Measure: Number; unit: parathyroid glands
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
parathyroid glands | 45 | 45

6. Secondary Outcome: Median Number of Parathyroid Glands Identified With NIRAF (PTeye Group Only)
Description: Median number of parathyroid glands identified with NIRAF, which was not seen with surgeon's naked eye during bilateral neck explorations (where the surgeon is looking for more than 1 parathyroid gland)
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Population: Only 4 participants had glands identified with NIRAF, which was not seen with surgeon's naked eye
Measure: Median (Full Range); unit: parathyroid glands
Arm/Group | Parathyroid Eye (PTeye)
Number analyzed (Participants) | 4
parathyroid glands | 1 [1 to 2]

7. Secondary Outcome: Median Number of Diseased Parathyroid Glands Identified Versus Preoperatively Localized Glands
Description: Median number of diseased parathyroid glands identified intra-operatively versus glands localized preoperatively using sestamibi, Computerized tomography (CT) or ultrasound
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Measure: Median (Full Range); unit: parathyroid glands
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
parathyroid glands
  Intra-operatively | 1 [1 to 2] | 1 [0 to 2]
  Localized pre-operatively | 1 [1 to 3] | 1 [1 to 3]

8. Secondary Outcome: Median Number of Intra-operative Parathyroid Hormone (PTH) Assays Sent
Description: The median number of intra-operative parathyroid hormone assays (per person) sent during the procedure to the lab
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Measure: Median (Full Range); unit: assays
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
assays | 5 [4 to 8] | 5 [4 to 12]

9. Secondary Outcome: Median Duration Taken to Identify First Parathyroid Gland
Description: Median duration in minutes taken to identify 1st parathyroid gland in PTx procedure - timed from skin incision to finding PG
Time Frame: During parathyroidectomy, up to 5 hours
Population: Data was not collected for one participant from each group
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 37 | 40
minutes | 38 [15 to 154] | 31 [11 to 184]

10. Secondary Outcome: Median Duration Taken to Identify Last Parathyroid Gland
Description: Median duration taken to identify last parathyroid gland in PTx procedure - timed from skin incision to finding the last PG
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Population: Data was not collected for one participant from each group
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 37 | 40
minutes | 48 [16 to 224] | 35 [11 to 184]

11. Secondary Outcome: Median Duration of Parathyroidectomy (PTx) Procedure
Description: Median duration of PTx procedure - timed from skin incision until the surgeon notifies the anesthesia team to awaken the patient in minutes
Time Frame: Up to 5 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
minutes | 87 [34 to 243] | 82 [26 to 296]

12. Secondary Outcome: Median Duration for Intraoperative Parathyroid Hormone (PTH) to Normalize
Description: Median time in minutes taken for PTH to attain cure criteria or normalize - timed from skin incision until the PTH levels drops > 50% of its baseline value and/or PTH drops < 65 pg/ml or 6.9 pmol/L
Time Frame: At the end of the parathyroidectomy, up to 5 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
minutes | 76 [27 to 243] | 66 [38 to 150]

13. Secondary Outcome: Median Number of Nights in the Hospital After Parathyroidectomy
Description: Median number of nights spent in the hospital post-surgery is defined as having spent <= 23 hours (0 nights) or > 23 hours (1 night) at the hospital for postoperative recovery after the surgical procedure. Participants who had surgery scheduled for later in the day will be counted as spending one night in the hospital due to the minimum required observation period post-surgery and followed institutional standards for discharge; discharged the next day. Participants who had surgery scheduled for earlier in the day were discharged on the same day of surgery.
Time Frame: 0-72 hours after PTx procedure
Measure: Median (Full Range); unit: number of nights
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 40
number of nights
  <= 23 hours | 0 [0 to 0] | 0 [0 to 0]
  > 23 hours | 1 [1 to 1] | 1 [1 to 1]

14. Secondary Outcome: Median Number of 'False Positive' Tissue Samples Excised by Surgeon
Description: The median number of tissues per person that were excised by surgeon assumed to be parathyroid tissue, but is later validated as non-parathyroid tissue (false positive) by histology
Time Frame: Up to 10 days after PTx procedure
Measure: Median (Full Range); unit: tissue samples
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
tissue samples | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Number of Participants With Reported Doctor Visits/Emergency Department Visits or Hospital Admissions
Description: Number of participants who required a doctor visit/emergency department visit and/or hospital admission due to persistent hypercalcemia and/or associated symptoms after the parathyroidectomy procedure will be categorized as binary (yes or no) if any follow-up visits or admissions occurred.
Time Frame: Up to 6 months after PTx procedure
Measure: Number; unit: participants
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
participants | 5 | 8

16. Secondary Outcome: Number of Participants Who Have Had Repeat Parathyroidectomy (PTx) Procedure
Description: Number of participants with an indication that repeat PTx procedure may need to be performed after the current procedure will be categorized as binary (yes or no)
Time Frame: From 6 - 12 months after PTx procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
Number analyzed (Participants) | 38 | 41
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Parathyroid Eye (PTeye) | Usual Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/38 | 5/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parathyroid Eye (PTeye) (N=38) | Usual Standard of Care (N=41)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Ovarian cancer
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps), Other - specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Myoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Benign hemangioma and benign angiolipoma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT05152927/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05152927/ICF_000.pdf